CLINICAL TRIAL: NCT06586268
Title: The SNORE-trial: Postoperative REM-Sleep Disturbance iN Obstructive Sleep-apnea Patients and the Relation With AH-index
Brief Title: The SNORE-trial: Analysis of Alterations in Sleep Stages Following Anesthesia and Their Relation to the Severity of Obstructive Sleep Apnea in the First 3 Nights After Surgery
Acronym: SNORE
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: VU University of Amsterdam (Other)
Responsible Party: Principal Investigator, Martin Rutten, MSc, MD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 2024.0163
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-09

CONDITIONS: Sleep Apnea Syndrome, Obstructive; Sleep Apnea Syndrome (OSAS)
Keywords: OSAS; OSA; obstructive sleep apnea; Post-surgical; post-anesthesia; REM sleep; PACU; AHI; Desaturations
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients scheduled for elective surgery with a diagnosis of obstructive sleep apnea (OSA): * Patients scheduled for elective surgery at the operating theatres of the AUMC with a diagnosis of OSA with or without treatment
  * Patients with continuous positive airway pressure (CPAP) or mandibular advancement device (MAD) are considered patients with treatment for OSA
  * Patients ≥ 18 years
  * Dutch or English speaking
  * Willing and able to sign consent for re-use of care data

SUMMARY:
The goal of this observational study is to learn about the relationship between sleep alterations following anesthesia and their relationship to a potential increase of obstructive sleep apnea (OSA) severity.

Our main question is: Is there an increased severity of OSA on the third post-operative night compared to the first post-operative night and does this have a relation with REM sleep?

Participants enrolled in this research are all diagnosed with OSA, with or without treament. All participants will be asked to wear a watchlike device called WATCHPAT to identify sleep paterns and register apneic (no breathing) and hypopneic (insufficient breathing) incidents. We ask our participants to wear this device for 8-10 hours a night when they are a sleep.

DETAILED DESCRIPTION:
The study is a prospective, observational, single center cohort study on electively scheduled adult surgical patients at the Amsterdam UMC, Amsterdam, The Netherlands.

Patients eligible for inclusion will be identified at the pre-operative screening at the outpatient clinic and contacted and included prior to the day of surgery.

Patients will sign an informed consent. Alternatively patients will be identified by an electronic algoritm which will analyse the next weeks elective surgery list. the algorithm analyzes for sleap apnea; in the patient problem list in their electronic patient file. Patients that have not been identified at the outpatient clinic will be able to be identified as eligible for inclusion via this route.

Measurement will start post-operatively at the recovery ward. All data will be registered with a non-invasive device, the WatchPAT (ZOLL medical). This device will measure apneic and hypopneic incidents, reported as apneu-hypopneu index (AHI) and vital signs such as blood pressure, heart rate and oxygen saturation. In addition the Watchpat will register REM-sleep via actigrapy. Other patient characteristics and demographics will be retrieved from the electronic patient file (EPIC).

These measurements will be started within 30 minutes of arriving at the recovery on the day of surgery continuing on into the first night at the PACU unit. On night 2 and 3 post-operatively participants will be asked to wear the device on the ward when going to sleep for the night. measurement period at the ward will be 8-10 hours.

For results on our primary outcome:

difference in mean of AHI and desaturations on night one compared to night three.

We aimed to detect a difference in mean of an AHI of 0.8 in a design with 3 repeated measurements when assuming a standard deviation of 2 and a very conservative between level correlation of 0. In order to detect a similar difference with a power of 80% and a significance level of 0.05, assuming a drop-out rate of 5%, we will need a sample size of 35 patients.

When patients are lost to follow up, or have incomplete measurements, defined as no functional data on sleep, AHI and desaturations in night 1 or night 3. Where a sleep time of 1,5 hours a night is minimally needed for complete calculations on AHI.

We will use descriptive statistics to present the characteristics of patients, using mean with standard deviation, or median with interquartile range for continuous data and as absolute frequencies with proportions for categorical data. The main outcome measure will be compared using a paired t-test. Correlations will be calculated using Pearsons correlation coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery at the operating theatres of the AUMC with a diagnosis of OSA with or without treatment with an expected admittance of a minimum of 3 days
* Patients with continuous positive airway pressure (CPAP) or mandibular advancement device (MAD) are considered patients with treatment for OSA
* Patients ≥ 18 years
* Dutch or English speaking
* Willing and able to sign consent for re-use of care data

Exclusion Criteria:

* Patients < 18 years
* Not speaking Dutch or English
* Patients who do not sign consent for re-use of care data
* Surgery scheduled in day case or with an expected discharge before the third night after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective surgery at the operating theatres of the AUMC with a diagnosis of OSA with or without treatment with an expected admittance of a minimum of 3 days
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
AHI and Desaturations on night one and three after surgery | from directly post operatively up untill the morning after the third night following surgery.
  To compare the AHI and desaturations on night one and night three after surgery

SECONDARY OUTCOMES:
Desaturations post operatively | The first six hours after surgery
  Assess the amount of patients with na increase of respiratory events (saturation <90%) later than 6 hours after surgery.
AHI directly post-operatively | directly post-operatively up untill the next morning (max 24 hours)
  compare the difference between AHI and desaturations in the first six hours after surgery to the first night after surgery.
Changes in total REM sleep | The first three nights following surgery
  Changes in total REM sleep comparing night 1,2 and 3.
Changes in AHI, REM-AHI and desaturations over time | Night one, two and three.
  To analyze the changes over time in AHI, REM-AHI, (respiratory events related tot REM-sleep cycle) and desaturations.
REM sleep and AHI | From directly post-operatively up untill the morning after the third night.
  Correlation between REM Sleep and respiratory events measured as AHI
Comparison of patients with treatment and patients without treatment | DIrectly post-operatively up untill the morning after night three
  Comparing AHI and desaturations between patients with either a MRA or CPAP treatment to those without any form of treatment or other treatment than MRA and CPAP.
Morfine and AHI/desaturations | from directly post-operatively to the morning after the third night.
  Compare respiratory events measured as AHI or desaturations compared to opioid consumption, measured as morphine equivalents.
  identifying different time-frames.
  * the first 6 hours after surgery
  * the first night after surgery (excluding the first six hours)
  * night 2 and night 3 after surgery.
  also identifying different modalities if applicable.
  * IV (patient controled and nurse controled)
  * oral

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Hermanides, Prof. Dr., Principal Investigator — AmsterdamUMC
Locations (2):
- Netherlands (2):
  - AmsterdamUMC, location AMC, Amsterdam, North Holland
  - Amsterdam UMC location VuMC, Amsterdam

IPD SHARING:
Plan to Share IPD: Yes
Study-protocol: will be available upon request SAP ,ICV, CSR will all be able on request. Data will be anonymized when data shared is patient specific.
  There is no analytical code involved in our study. therefore this will not be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Study protocol, ICF (standard model) with SAP are available upon request as of now. (september 2024) Data will be available until 5 year after publishing.
Access Criteria: Only the researchteam will have direct acces to the researchdata and specific patient data.
  External requests will be evaluated by the principal investigator